CLINICAL TRIAL: NCT05628233
Title: A Phase IIa, Multicenter, Randomized, Controlled, Open Label Study to Evaluate the Efficacy of SENS-401 to Prevent the Ototoxicity Induced by Cisplatin in Adult Subjects With a Neoplastic Disease
Brief Title: SENS-401 to Prevent the Ototoxicity Induced by Cisplatin in Adult Subjects With a Neoplastic Disease
Acronym: NOTOXIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SENS-401-202
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss Ototoxic
MeSH Terms: interventions — SENS-401

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Arm A (control arm) (No Intervention): Subjects receiving cisplatin-based chemotherapy without receiving SENS-401. This control arm will provide natural history data, particularly the incidence and the time to onset of hearing impairment due to ototoxicity.
- Study Arm B (treatment arm) (Experimental): Subjects receiving 43.5 mg of oral SENS-401 b.i.d for up to 23 weeks. This arm will provide data on the potential protective effects of SENS-401 on cisplatin induced ototoxicity.
  Interventions: Drug: SENS-401 (R-Azasetron Besylate)

INTERVENTIONS:
Drug: SENS-401 (R-Azasetron Besylate) — Patients will receive SENS-401 ((R)-azasetron besylate) B.I.D. up to 23 weeks: 1 week prior to the initiation of the cisplatin treatment, during the whole duration of the chemotherapy treatment (estimated to last up to 18 weeks) and 4 weeks after stopping chemotherapy.
  Arms: Study Arm B (treatment arm)

SUMMARY:
This study is intended to evaluate the ability of SENS-401 to prevent the ototoxicity induced by cisplatin in subjects with a neoplastic disease. It is a multicenter, randomized, controlled, two-arm, open-label efficacy and safety study in adults with neoplastic disease requiring treatment with cisplatin as part of the chemotherapy protocol plan.

DETAILED DESCRIPTION:
This study is intended to evaluate the ability of SENS-401 to prevent the ototoxicity induced by cisplatin in subjects with a neoplastic disease. It is a multicenter, randomized, controlled, two-arm, open-label efficacy and safety study in adults with neoplastic disease requiring treatment with cisplatin as part of the chemotherapy protocol plan. Cisplatin treatment per chemotherapy protocol must be given at a cumulative dose high enough to significantly increase the iatrogenic likelihood of ototoxicity (unit cisplatin dose of at least 70 mg/m2 and cumulative cisplatin dose of at least 210 mg/m²). If all the eligibility criteria are met, subjects will be randomized to one of two study arms as follows:

* Study Arm A (control arm): Subjects receiving cisplatin-based chemotherapy without receiving SENS-401. This control arm will provide natural history data, particularly the incidence and the time to onset of hearing impairment due to ototoxicity.
* Study Arm B: Subjects receiving 43.5 mg of oral SENS-401 b.i.d for up to 23 weeks: 1 week prior to the initiation of the cisplatin treatment, during the whole duration of the chemotherapy treatment (estimated to last up to 18 weeks) and 4 weeks after stopping chemotherapy. This arm will provide data on the potential protective effects of SENS-401 on cisplatin induced ototoxicity.

All subjects will be followed up to 12 weeks after the completion of the cisplatin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the ICF.
2. Neoplastic subject that regardless of participation in this study is planned to be treated with a chemotherapy that includes a dose of cisplatin of at least 70 mg/m² per cycle and a cumulative dose of cisplatin of at least 210 mg/m².

Exclusion Criteria:

1. Any condition or past medical history that, in the opinion of the Investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study.
2. A congenital or hereditary disease known to decrease hearing function.
3. Any medical history affecting the middle ear function such as chronic otitis, cholesteatoma, or tympanic membrane perforation.
4. Any inner ear disease that is likely to decrease hearing function according to the Investigator's judgment (e.g, herpes zoster oticus; Meniere's disease; purulent labyrinthitis; vestibular schwannoma).
5. Having a history of sudden sensory neural hearing loss.
6. Having a fluctuating hearing loss (e.g, due to Meniere's disease, vestibular aqueduct syndrome, or autoimmune inner ear disease).
7. History of head trauma with hearing loss.
8. History of meningitis.
9. Having received concomitant treatment known or suspected to induce an ototoxicity within 6 months prior to Screening (i.e, aminoglycosides, loop diuretics, quinine) and any other treatments listed in Appendix 5. Previous treatment with a platinum treatment should be considered as an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
SENS-401 efficacy assessment with change from baseline of the average of the hearing threshold 4 weeks after the completion of cisplatin treatment | 23 weeks
  Change from baseline of the average of the hearing threshold of 3 contiguous hearing frequencies assessed with a 0.5-12.5 kHz audiogram 4 weeks after the completion of the last cisplatin treatment in each ear of each subject.

SECONDARY OUTCOMES:
SENS-401 efficacy assessment with change from baseline of the average of the hearing threshold 12 weeks after the completion of cisplatin treatment. | 31 weeks
  Change from baseline of the average of the hearing threshold of 3 contiguous hearing frequencies assessed with a 0.5-12.5 kHz audiogram 12 weeks after the completion of the last cisplatin treatment in each ear of each subject.
SENS-401 efficacy assessment with change from baseline in the distribution of hearing loss severity 4 weeks after the completion of cisplatin treatment | 23 weeks
  Change from baseline in the distribution of hearing loss severity at 4 weeks after the completion of cisplatin treatment. The severity of the hearing loss being based on the CTCAE (version 5.0).
SENS-401 efficacy assessment with change from baseline in the distribution of hearing 12 weeks after the completion of cisplatin treatment | 31 weeks
  Change from baseline in the distribution of hearing loss severity at 12 weeks after the completion of cisplatin treatment. The severity of the hearing loss being based on the CTCAE (version 5.0).
SENS-401 efficacy assessment with change from baseline in speech discrimination test score 4 weeks after the completion of cisplatin treatment. | 23 weeks
  Change from baseline in speech discrimination test score (assessed in noise and in quiet) 4 weeks after the completion of the cisplatin treatment.
SENS-401 efficacy assessment with change from baseline in speech discrimination test score 12 weeks after the completion of cisplatin treatment | 31 weeks
  Change from baseline in speech discrimination test score (assessed in noise and in quiet) 12 weeks after the completion of the cisplatin treatment.
SENS-401 efficacy assessment with change from baseline in Tinnitus Handicap Inventory (THI) Questionnaire score 4 weeks after the completion of cisplatin treatment. | 23 weeks
  Change from baseline in Tinnitus Handicap Inventory (THI) Questionnaire score, 4 weeks after the completion of the cisplatin treatment.
SENS-401 efficacy assessment with change from baseline in Tinnitus Handicap Inventory (THI) Questionnaire score 12 weeks after the completion of cisplatin treatment | 31 weeks
  Change from baseline in Tinnitus Handicap Inventory (THI) Questionnaire score,12 weeks after the completion of the cisplatin treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No